CLINICAL TRIAL: NCT01216059
Title: The Use of Text Messages to Improve Adherence to Health Maintenance Behaviors in Adolescents With Atopic Dermatitis
Brief Title: Text Messaging and Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Professor and Chair of Department of Dermatology, Professor of Pediatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU29486
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Atopic Dermatitis
Keywords: adherence; text message; reminder; adolescents
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Subjects will receive daily text message reminder about their treatment for atopic dermatitis during the 6 weeks of the study.
  Interventions: Procedure: Text message to cell phone
- Control Group (No Intervention): Subjects will receive a weekly text message reminder about pop-culture, sports or weather.

INTERVENTIONS:
Procedure: Text message to cell phone — Subjects will receive a daily text message reminder about their treatment for atopic dermatitis during the 6 weeks of the study
  Arms: Intervention group

SUMMARY:
Atopic dermatitis is a common problem faced by patients of all ages and backgrounds. Treatment regimens and specific therapies may be time consuming and multiple studies have documented a parallel decrease in compliance as time after an office visit increases. The adolescent population is an extremely challenging sub-group of patients in terms of complying with a treatment regimen. Not only are they striving for independence and thus lacking supervision of a regimen by a parent, but their complex thinking skills are immature, leading to forgetful behavior. By introducing a reminder system for these vulnerable patients that is easily incorporated into their daily lives, the investigators propose that patients will have better compliance at applying their medication and thus improving their atopic dermatitis. Text-messaging via cell phones has become very popular among teenagers and adults and provides a non-obtrusive method of sending a treatment reminder.

DETAILED DESCRIPTION:
We propose to conduct a randomized, controlled 6-week trial to evaluate the impact of a text message-based reminder program on adherence to health maintenance behaviors among adolescents diagnosed with Atopic Dermatitis. After obtaining informed consent, subjects will be randomized into either an intervention or control group. Subjects in the intervention group will receive a daily text message with a tailored message regarding atopic dermatitis, while control group subjects will receive a weekly text message with information on local weather, sport or news without any reference to atopic dermatitis. Of note, the decision to send a weekly text message to the control group reflects the expectation that a message will be sent, although the frequency and content of the message will not be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 inclusive
* Capable of giving informed consent/assent. Of note, all subjects will sign an assent form and parents will sign a parent consent form.
* Diagnosed with Atopic Dermatitis by a physician (self report)
* IGA score fo 2 or greater
* Currently using at least one prescribed topical therapy for atopic dermatitis
* Have a mobile phone capable of receiving text messages
* Able to retrieve text messages from mobile phone
* Able to adhere to study visit schedule and other protocol requirements.

Exclusion Criteria:

* Younger than 10 years of age or 18 years and older at the time of enrollment
* No diagnosis of atopic dermatitis by a physician
* IGA score of 0 or 1
* Currently on no prescribed topical treatment for atopic dermatitis
* UV therapy or climatotherapy is a part of treatment for atopic dermatitis
* Does not have a mobile phone capable of receiving text messages
* Unable to retrieve text message
* Non-English speaking individuals (text messages are in English)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in self reported medication adherence | 6 weeks
  We will assess the difference in number of missed doses of topical medication in the control group (weekly unrelated text message) and the intervention group (daily eczema-related text message group). All subjects will record missed doses via calendars (diaries). Those in the intervention group will be able to text on a weekly basis the number of days they forgot their medication that week.
Change in quality of life | 6 weeks

SECONDARY OUTCOMES:
Change in AD knowledge score | 6 weeks
Change in health maintenance behaviors | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois